CLINICAL TRIAL: NCT04156880
Title: Breast Cancer Screening With Mammography: Diagnostic Assessment of an Artificial
Brief Title: Artificial Intelligence in Mammography-Based Breast Cancer Screening
Status: Withdrawn | Type: Observational
Why Stopped: the collaborating party of AI system withdraw their study due to change of company policy in year of COVID-19 pandemic
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: IBM China/Hong Kong Limited (Unknown)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Other Study IDs: 2019.629
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: mammography; artificial intelligence; deep learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mammography — standard mammography including craniocaudal (CC) and mediolateral oblique (MLO) views

SUMMARY:
Breast cancer (BC) is the most common cancer among women in worldwide and the second leading cause of cancer-related death.

As the corner stone of BC screening, mammography is recognized as one of useful imaging modalities to reduce BC mortality, by virtue of early detection of BC. However, mammography interpretation is inherently subjective assessment, and prone to overdiagnosis.

In recent years, artificial intelligence (AI)-Computer Aided Diagnosis (CAD) systems, characterized by embedded deep-learning algorithms, have entered into the field of BC screening as an aid for radiologist, with purpose to optimize conventional CAD system with weakness of hand-crafted features extraction. For now, stand-alone performance of novel AI-CAD tools have demonstrated promising accuracy and efficiency in BC diagnosis, largely attributed to utilization of convolution neural network(CNNs), and some of them have already achieved radiologist-like level. On the other hand, radiologists' performance on BC screening has shown to be enhanced, by leveraging AI-CAD system as decision support tool. As increasing implementation of commercial AI-CAD system, robust evaluation of its usefulness and cost-effectiveness in clinical circumstances should be undertaken in scenarios mimicking real life before broad adoption, like other emerging and promising technologies. This requires to validate AI-CAD systems in BC screening on multiple, diverse and representative datasets and also to estimate the interface between reader and system. This proposed study seeks to investigate the breast cancer diagnostic performance of AI-CAD system used for reading mammograms. In this work, we will employ a commercially available AI-CAD tool based on deep-learning algorithms (IBM Watson Imaging AI Solution) to identify and characterize the suspicious breast lesions on mammograms. The potential cancer lesions can be labeled and their mammographic features and malignancy probability will be automatically reported. After AI post-processing, we shall further carry out statistical analysis to determine the accuracy of AI-CAD system for BC risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Women who had undergone standard mammography including craniocaudal (CC) and mediolateral oblique (MLO) views..
* Histopathology-proven diagnosis is available for patients with breast malignancy, including invasive breast cancer, carcinoma in situ, and borderline lesion et al.
* As reference standard of benign nature, results from pathology or clinical long-term follow-up (>=2 years) examinations are available for cases without breast malignancy.

Exclusion Criteria:

* Patients with concurring lesions on mammograms that may influence subsequent AI post-process.
* Patients without available pathologic diagnosis or long-term follow-up (>=2 years) examinations.
* Patients who had undergone breast surgical intervention (e.g. lumpectomy and mammoplasty) prior to first mammography.
* Patients diagnosed with other kinds of malignancy, concurrent with metastasis or infiltration/invasion to breast.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is a single institutional retrospective cohort study of patients with mammographic examinations. All patients' data will be retrieved via the electronic patient database of our institution. Patient demographics, imaging and histological data, disease and treatment history will be recorded, including age at onset, details of chemotherapy, time interval of metastasis from diagnosis, surgery for the primary tumor, the length of survival, clinical outcome and so on.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
area under curve (AUC) | 3 years
  area under receiver operating characteristic (ROC) curve in percentage (%)
accuracy | 3 years
  proportion of true results(both true positives and true negatives) among whole instances
sensitivity | 3 years
  true positive rate in percentage(%) derived by ROC analysis
specificity | 3 years
  true negative rate in percentage (%) derived by ROC analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong